CLINICAL TRIAL: NCT03505593
Title: A Feasibility Study to Evaluate the Clinical Safety of ENvizion Medical™ Enteral Feeding Tube Placement Using the ENvizion Medical™ ENVUE™ System in Patients
Brief Title: Feasibility Study to Evaluate Safety of ENvizion Medical™ ENVUE™ System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Envizion Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NUTRI002
Record Dates: First submitted 2018-04-09; First posted 2018-04-23 (Actual); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-03

CONDITIONS: Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EFT placement using ENVUE System (Experimental): Placement of the ENvizion Medical™ Enteral Feeding Tube (EFT) in the stomach or small intestine of adult patients who require feedings via the oro/ nasoenteric route, using the ENVUE™ System.
  Interventions: Device: ENVUE System

INTERVENTIONS:
Device: ENVUE System — The ENvizion Medical™ ENVUE™ System is designed to aid qualified operators in the placement of the ENvizion Medical™ Enteral Feeding Tube™ into the stomach or small intestine.

SUMMARY:
This is a single center, non-randomized feasibility clinical evaluation that is designed to affirm the safety of the ENVUE™ System guidance during the placement of the ENvizion Medical™ enteral feeding tubes.

DETAILED DESCRIPTION:
Enteral nutrition is the preferred route for the provision of nutritional support in most critical ill patients with functional gastrointestinal tract. Achieving early enteral nutrition (EN) in critically ill patients is associated with fewer major complications, reduced mortality and length of hospital stay, and significant cost savings. It is estimated that approximately 1.2 million feeding tubes are placed blindly each year in the United States alone. Despite the obvious advantages of the enteral tube feeding, inadvertent placement of Enteral Feeding Tube (EFT) into the airway is relatively common and can result in significant pulmonary injury including pneumothorax and pneumonia. Airway misplacement occurs in 1.2- 4 % of blind EFT insertions, with 0.2 to 1.2% of all the feeding tube placements cause pulmonary complications to patients. The gold standard for detecting inadvertent placement of a feeding tube in the lungs is radiography. However, because of its cost, possible delay of feedings while waiting for radiography, and risk for radiation exposure, clinicians continue to seek for alternative methods to confirm correct placement.

All the above mentioned, emphasizes the fact that safe and effective delivery of nasoenteral tube feedings requires assurance that the feeding tube tip is in a proper position. The ENVUE™ System is an electromagnetic tracking system which tracks the path of the feeding tube during placement. The benefit of the system when EFT is misdirected into the pulmonary system is a real-time visual tracing, which may prompt users to withdraw the tube and reinsert it.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >21 years of age
* Patients must require placement of an enteral feeding tube
* Patients have an endotracheal tube, OR Do not have an endotracheal tube but are sedated (RASS score of -2 or less) and/or obtunded (Glasgow Coma scale of 9-12)
* Patients or legal authorized representative must be able to understand and adhere to all protocol procedures and be willing and able to provide written informed consent

Exclusion Criteria:

* Patients must not have a history of:

  * Esophageal varices or ulcers
  * Upper airway obstruction
  * Upper GI stenosis or obstruction
  * Trauma involving sinuses, nares face or neck that would prevent nasogastric (NG) or oral tube insertion
  * Deformities of the sinus cavities and/or skull base
  * Esophageal cancer or neoplasm
* Patients must not have a significant concomitant illness that would adversely affect their participation in the study
* Female patients who are pregnant or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Jacobson, MD, Principal Investigator — St.Vincent Hospital and Health Care Center, Inc.
Locations (1):
- St.Vincent Hospital and Health Care Center, Inc., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 48 enrolled participants, 46 met inclusion/ exclusion criteria and underwent a tube placement attempt. From these 46 participants, 43 completed a successful tube placement.
Period: Overall Study
Arm/Group | EFT Placement Using ENVUE System
Started | 48
Completed | 43
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Died before procedure | 1
Not completed — Anatomical abnormality | 1
Not completed — Unable to pass through esophagus | 1
Not completed — Obstruction by Endotracheal tube | 1

BASELINE CHARACTERISTICS:
Arm/Group | EFT Placement Using ENVUE System
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 67 [28 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3
  White | 40
Region of Enrollment [Number; unit: participants]
  United States | 43
Sedated [Count of Participants; unit: Participants] | 0
Obtunded [Count of Participants; unit: Participants] | 5
Endotracheal Tube [Count of Participants; unit: Participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successfully Placed Enteral Feeding Tube
Description: Enteral tube (EFT) can be placed in the correct anatomical position without occurrence of guidance-related adverse events.
  Procedure success was evaluated by comparing tube tip location according to the ENVUE System and abdominal and/or thoracic X-Ray.
  Guidance-related AEs were evaluated through the documentation of any guidance-related serious adverse events (SAE) or adverse events (AE) occurring during a subject's participation in the study.
Time Frame: During procedure visit
Population: Subjects who underwent a successful feeding tube placement using the ENvue system
Measure: Count of Participants; unit: Participants
Arm/Group | EFT Placement Using ENVUE System
Number analyzed (Participants) | 43
Participants | 43

2. Secondary Outcome: Total Number of Placement Attempts
Description: Number of placement attempts was evaluated by number of replacement and repositioning events, as defined below:
  * Replacement: Complete removal of the tube from the patient or retraction above the level of the pharynx followed by reinsertion
  * Repositioning: Changing position of tube without complete removal of the tube
Time Frame: During procedure visit
Population: 43 subjects underwent a successful feeding tube placement using the ENvue system. In total, 44 tubes were successfully placed- 1 subject pulled the tube out and a new tube was placed instead
Measure: Number; unit: Number of placement attempts
Arm/Group | EFT Placement Using ENVUE System
Number analyzed (Participants) | 43
Number of placement attempts | 49

3. Secondary Outcome: Number of Retrograde Tube Migration Events
Description: Tube Migration was defined as: Retrograde migration from desired placement position.
Time Frame: During follow-up visit (20-48 hours post tube placement)
Population: 43 subjects underwent a successful feeding tube placement using the ENvue system.
  Of the Forty- three (43) subjects that completed a successful placement procedure, thirty-six (36) subjects underwent a successful tube tip position check at follow-up visit.
Measure: Number; unit: Number of tube retrograde migration
Arm/Group | EFT Placement Using ENVUE System
Number analyzed (Participants) | 36
Number of tube retrograde migration | 3

ADVERSE EVENTS:
Time Frame: From the participant's tube placement procedure (day 0) to the end of of the follow-up visit (20-48 hours post tube placement)
Description: Analysis was performed on all enrolled subjects (48 subjects)
Arm/Group | EFT Placement Using ENVUE System
All-Cause Mortality (participants affected / at risk) | 1/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 1/48
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EFT Placement Using ENVUE System (N=48)
Enteral feeding tube distal tip deattachement (Product Issues) | 1 (1) — Between the feeding tube placement procedure and follow-up visit, the tip of the tube became detached from the rest of the tube. The tip tube left the patient's body in a natural manner (during bowel movements).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Twelve months following the completion of the study, Investigator may publish the results of the study. Investigator shall provide sponsor advanced copies of any proposed publication sixty days prior to planned publication Sponsor will have sixty days to review the proposed publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT03505593/Prot_SAP_000.pdf